CLINICAL TRIAL: NCT06801496
Title: The Application of Gastric Bypass Stents in Patients with Weight Regain After Laparoscopic Sleeve Gastrectomy：a Feasibility Study
Acronym: DJBL for LSG
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hua Meng, irector of the General Surgery Department & Obesity and Metabolic Disease Center of China-Japan Friendship Hospital, China-Japan Friendship Hospital
Other Study IDs: 2023-KY-125
Record Dates: First submitted 2025-01-25; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-06

CONDITIONS: Obesity and Obesity-related Medical Conditions; Weight Regain
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is based on the National Center for Integrated Traditional Chinese and Western Medicine, utilizing the centralized advantages of our department and integrating multiple disciplines (general surgery, endocrinology, nutrition, sports, and traditional Chinese medicine). It focuses on the effectiveness of gastric bypass stents in treating patients with postoperative obesity after laparoscopic sleeve gastrectomy, as well as in patients with simple obesity. This will improve the prognosis of patients and reduce the medical burden.

ELIGIBILITY:
Inclusion Criteria:

* 1、For those with simple obesity, BMI ≥ 32.5, or 27.5 ≤ BMI < 32.5, who have difficulty controlling their condition with lifestyle modifications and medical treatment, and who meet at least two criteria for metabolic syndrome components, or have comorbidities.

  2、For those with simple obesity, 27.5 ≤ BMI < 32.5, and with male waist circumference ≥ 90 cm, female waist circumference ≥ 85 cm, and imaging studies suggesting central obesity.

  3、For those with type 2 diabetes, BMI ≥ 27.5, who still have some residual insulin secretion capacity.

Exclusion Criteria:

* 1、Non-obese type 1 diabetes; 2、Those for whom the purpose of treatment is T2DM, but whose pancreatic beta-cell function is largely lost, with a BMI < 25.0; 3、Age < 16 years or age > 65 years; 4、Pregnant women with diabetes and patients with certain special types of diabetes; 5、Those with a cognitive disorder or immature intelligence, and who cannot control their behavior; 6、Those whose expectations for the surgery are not realistic; 7、Those unwilling to assume the risks of potential surgical complications; 8、Those unable to comply with postoperative dietary and lifestyle changes, showing poor compliance; 9、Those in poor general health, who are unable to tolerate general anesthesia or surgery.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals planning to undergo bariatric surgery in China-Japan Friendship Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
weight | Before bariatric surgery, 1 month after surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing, Beijing, China